CLINICAL TRIAL: NCT00514956
Title: Effect of Emotional Freedom Technique and Diaphragmatic Breathing on PTSD
Brief Title: Effect of Emotional Freedom Technique and Diaphragmatic Breathing on Post Traumatic Stress Disorder (PTSD)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Soul Medicine Institute (Other)
Responsible Party: Dawson Church, Executive Director, Soul Medicine Institute
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: PTSD-ACEP-SMI-MU-1
Record Dates: First submitted 2007-08-08; First posted 2007-08-10 (Estimated); Last update posted 2009-09-22 (Estimated); Status verified 2009-09

CONDITIONS: Stress Disorders, Post-Traumatic
Keywords: Post-Traumatic Stress Syndrome (PTSD)
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Combat Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: Emotional Freedom Techniques (EFT)

SUMMARY:
A great many soldiers are returning from Iraq and Afghanistan with symptoms of Post Traumatic Stress Disorder (PTSD). Clinical experience with many people has shown the effectiveness of the techniques of Energy Psychology for rapidly alleviating PTSD symptoms. The study proposes to determine whether a very brief course of treatment (3 sessions) with a common form of Energy Psychology called Emotional Freedom Techniques (EFT) has an effect on the stress biochemistry of subjects, by measuring their levels of stress hormones (cortisol, DHEA) before and after treatment.

DETAILED DESCRIPTION:
The Purpose of the Research: The purpose of this study is to test the effectiveness of Emotional Freedom Technique (EFT) versus Diaphragmatic Breathing in Reducing Post Traumatic Stress Disorders.

The Scientific or Scholarly Rationale: Clinical experience and anecdotal reports have demonstrated EFT to be effective for a wide range of behavioral disorders, including PTSD. However with the exception of several studies demonstrating the efficacy of EFT for the treatment of simple phobias, there have been no formal research studies in this area. It is the intention of this study to extend the phobia studies to the area of PTSD, and to determine what other conditions EFT might be effective in treating. Another intention of this study is to see whether, and to what degree, changes in psychological functioning (as measure by the PAI and TSI) are reflected in physiological markers such as HRV (Heart Rate Variability) and levels of cortisol and DHEA.

The Procedures to be Performed: Approximately 8 to 10 subjects would be randomly designated to either the experimental or Diaphragmatic Breathing control groups. There will be 4-5 subjects in the EFT experimental group and 4-5 subjects in the control Diaphragmatic Breathing group.

ELIGIBILITY:
Inclusion Criteria:

* PTSD
* Recent Service in Afghanistan or Iraq
* Good Health History

Exclusion Criteria:

* Illegal Drug Use
* Recent Physical Trauma
* Head injuries, concussions, amputees
* Mental health issues prior to entering military service

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2007-09; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Change in baseline cortisol and DHEA production | Six months

SECONDARY OUTCOMES:
Changes in scores on Trauma Assessment Inventory and other instruments normed for trauma | Six months

CONTACTS AND LOCATIONS:
Overall Officials: Dawson Church, PhD, Study Director — Soul Medicine Institute
Locations (2):
- United States (2):
  - Marshall University Medical School, Charleston, West Virginia
  - Marshall University, Joan Edwards School of Medicine, Huntington, West Virginia

REFERENCES:
- [Result] Church, D., Geronilla, L., & Dinter, I. (2009) Psychological symptom change in veterans after six sessions of Emotional Freedom Techniques (EFT). International Journal of Healing and Caring, January, 9:1.
- See also: Web site to connect veterans to assistance using study protocol, and enrollment option for larger followup study. — http://www.StressProject.org